CLINICAL TRIAL: NCT01308606
Title: A Phase I, Open-label, Randomized, Single-dose, 2-panel, Crossover Trial in Healthy Subjects to Assess the Relative Bioavailability of TMC435 HPMC Capsule Compared to the TMC435 Gelatin Capsule and to Assess the Effect of Different Meal Types on the Bioavailability of Both Formulations
Brief Title: TMC435-TiDP16-C116 - Relative Bioavailability and Food Effect Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tibotec Pharmaceuticals, Ireland (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR015940; TMC435-TiDP16-C116
Record Dates: First submitted 2011-03-03; First posted 2011-03-04 (Estimated); Last update posted 2012-10-11 (Estimated); Status verified 2012-10

CONDITIONS: Hepatitis C
Keywords: TMC435-TiDP16-C116; TMC435-C116; TMC435; HCV; Hepatitis C; Hep C; healthy volunteers
MeSH Terms: conditions — Hepatitis C | interventions — Gelatin

ARMS (5):
- 001 (Experimental): TMC435 gelatin capsule Single intake of one 150-mg capsule without food
  Interventions: Drug: TMC435 gelatin capsule
- 002 (Experimental): TMC435 HPMC capsule Single intake of one 150-mg capsule without food
  Interventions: Drug: TMC435 HPMC capsule
- 003 (Experimental): TMC435 HPMC or gelatin capsule Single intake of one 150-mg capsule without food
  Interventions: Drug: TMC435 HPMC or gelatin capsule
- 004 (Experimental): TMC435 HPMC or gelatin capsule Single intake of one 150-mg capsule after standardized breakfast
  Interventions: Drug: TMC435 HPMC or gelatin capsule
- 005 (Experimental): TMC435 HPMC or gelatin capsule Single intake of one 150-mg capsule after high-fat breakfast
  Interventions: Drug: TMC435 HPMC or gelatin capsule

INTERVENTIONS:
Drug: TMC435 HPMC capsule — Single intake of one 150-mg capsule without food
  Arms: 002
Drug: TMC435 HPMC or gelatin capsule — Single intake of one 150-mg capsule after high-fat breakfast
  Arms: 005
Drug: TMC435 HPMC or gelatin capsule — Single intake of one 150-mg capsule without food
  Arms: 003
Drug: TMC435 HPMC or gelatin capsule — Single intake of one 150-mg capsule after standardized breakfast
  Arms: 004
Drug: TMC435 gelatin capsule — Single intake of one 150-mg capsule without food
  Arms: 001

SUMMARY:
The purpose of this study is to compare absorption of TMC435 formulated as 2 different types of capsules. After that, the absorption of one chosen TMC435 capsule will be compared when taken under fasting conditions or together with a standard or a high-fat meal. This will be done in healthy volunteers.

DETAILED DESCRIPTION:
This is an open-label, randomized, single-dose, crossover trial in healthy volunteers. Crossover means that participants may receive different interventions sequentially during the trial. Randomized means that you will be assigned to a treatment sequence by chance, like flipping a coin. Open-label means that you and your physician will know what treatment you will receive. The study will consist of 3 phases: a screening phase, a treatment phase and a follow-up phase. Total study duration for an individual participant will be up to 6 or 7 weeks. Once found eligible after the screening phase, participants will take part in one of the two parts of the treatment phase. In the first part, a group of 24 participants will receive two treatment sessions, A and B. The order in which the treatments are given will be determined by chance. Treatment A is a single dose of TMC345 as one formulation (1 capsule). Treatment B is a single dose of TMC435 as another formulation (1 other type of capsule). Both treatments will be taken without food. In between the 2 sessions, there will be at least 7 days. In the second part, another group of 24 participants will receive 3 treatment sessions, C, D, and E. The order in which these treatments are given will be determined by chance. All 3 treatments will consist of a single dose of TMC435 as one of the 2 formulations given in the first part. In Treatment C this will be given without food, in Treatment D with a standardized breakfast and in Treatment E with a high-fat breakfast. In between the sessions, there will be at least 7 days. For all treatment sessions, participants will enter the study center the day before dosing and will remain there until the evening of the day after. The 3 following mornings, participants will come back to the study center. Five to 7 days after dosing, participants will have a last follow-up visit at the study center (follow-up phase). During the study, safety will be monitored, and during the treatment phase, at specified timepoints, blood samples will be taken for pharmacokinetic evalutions (effect of the body on the drug). In every treatment session, a single oral 150 mg TMC435 capsule will be given. One formulation will be a gelatin capsule. The other formulation will be a hydroxypropylmethylcellulose (HPMC) capsule.

ELIGIBILITY:
Inclusion Criteria:

* Non-smokers for at least 3 months prior to screening
* Have a body mass index of 18.0 to 30.0 kg per square meter
* Be healthy on the basis of physical examination, medical history, vital signs, and clinical laboratory tests performed at screening

Exclusion Criteria:

* Use of disallowed therapies, including over-the-counter products and dietary supplements
* Having previously participated in a multiple-dose trial or more than 3 single-dose trials with TMC435
* Received an investigational drug or used an investigational medical device within 90 days before the planned start of treatment
* History or evidence of current use of alcohol, barbiturate, amphetamine, recreational, or narcotic drug use

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2011-03; Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Absorption of TMC435 following administration of the HPMC capsule and of the gelatin capsule | Over 72 hours for every treatment session
Absorption of TMC435 following administration of the HPMC or gelatin capsule in the fed (following different meal types) and fasted state | Over 72 hours for every treatment session

SECONDARY OUTCOMES:
Number of participants with adverse events and the severity of adverse events | During maximum 7 weeks
Percentage of abnormal values for laboratory parameters | Up to maximum 7 weeks
Observed values and changes from baseline of cardiovascular variables | Up to maximum 7 weeks
Evaluation of pulse and blood pressure values, based on changes from baseline and the percentage of participants with values beyond clinically important limits | Up to maximum 7 weeks
Physical examination findings and changes from baseline. | Up to maximum 7 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Tibotec Pharmaceuticals Clinical Trial, Study Director — Tibotec Pharmaceutical Limited